CLINICAL TRIAL: NCT02734563
Title: Collagen Alterations in Patients With Abdominal Wall Hernias
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Lars Nannestad Jorgensen, Professor, MD, Bispebjerg Hospital
Other Study IDs: H.A-2009-045
Record Dates: First submitted 2016-04-01; First posted 2016-04-12 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Hernia, Abdominal
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Multiple hernia group: Males undergoing at least three repairs of abdominal wall hernias at three different anatomic locations. Collagen turnover is analysed.
  Interventions: Other: Collagen turnover
- Control group: Males without any history or presence of hernias
  Interventions: Other: Collagen turnover

INTERVENTIONS:
Other: Collagen turnover — Type IV and V collagen synthesis and breakdown

SUMMARY:
The aim of this study was to evaluate collagen turnover in patients with multiple hernias

DETAILED DESCRIPTION:
Venous blood was collected and markers for type IV and V collagen synthesis and breakdown was measured

ELIGIBILITY:
Inclusion Criteria:

* patients with a history of three hernia repairs (multiple hernia group)
* patients without any history or presence of hernias (control group)

Exclusion Criteria:

* connective tissue disorder (Ehlers-Danloss/Marfan)
* presence of hernia upon clinical examination (control group)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males with multiple hernias wer identified from the Danish Hernia Database. The control group were recruited from hospital staff.
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Type IV and V collagen synthesis and breakdown | 3 months
  Products from type IV and V collagen synthesis and breakdown are measured in serum. with ELISA from Nordic Bioscience A/S, Herlev, Denmark. Specifically, the biomarker for type IV collagen synthesis (P4NP) and breakdown (C4M), and for type V collagen synthesis (P5CP) and breakdown (C5M) was measured. The concentration unit for all parameters is ng/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Lars N Jorgensen, MD, Principal Investigator — Bispebjerg Hospital, Dept. of Surgery
Locations (1):
- Bispebjerg Hospital, Copenhagen, NV, Denmark

IPD SHARING:
Plan to Share IPD: No